CLINICAL TRIAL: NCT01354340
Title: Dose Effect of Limicol on (LDL)-Cholesterol Levels in Moderate Hypercholesterolaemia
Brief Title: Dose Effect of Limicol on (LDL)-Cholesterol Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lescuyer Laboratory (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011-A00145-36
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Hypercholesterolaemia
Keywords: Cholesterol; LDL-cholesterol; Coronary artery disease; Red yeast rice; Plants extract; Cholesterol excess; Delivery of Health Care
MeSH Terms: conditions — Hypercholesterolemia; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Limicol simple dose (Experimental)
  Interventions: Dietary Supplement: Limicol
- Limicol double doses (Experimental)
  Interventions: Dietary Supplement: Limicol
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Limicol — 3 tablets (Limicol) + 3 tablets (Placebo) / day during 1 month and follow-up 1 month without treatment
  Arms: Limicol simple dose
Dietary Supplement: Limicol — 6 tablets (Limicol) / day during 1 month and follow-up 1 month without treatment
  Arms: Limicol double doses
Other: Placebo — 6 tablets (Placebo) / day during 1 month and follow-up 1 month without treatment
  Arms: Placebo

SUMMARY:
The principal objective of this study is to investigate the dose-effect of the Limicol food supplement on LDL-cholesterol level in moderate hypercholesterolaemia subjects.

ELIGIBILITY:
Inclusion Criteria:

* About 18 to 65 years (inclusive).
* Subject has a stable weight for at least three months before the start of the study.
* Subject able and willing to comply with the protocol and agreeing to give their consent in writing.
* Subject affiliated with a social security scheme.
* Subject willing to be included in the national register of volunteers who lend themselves to biomedical research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in blood LDL-cholesterol levels after 4 weeks of supplementation (limicol double dose group versus placebo group) | 4 weeks after baseline

SECONDARY OUTCOMES:
Change from Baseline in blood LDL-cholesterol levels after 4 weeks of supplementation (limicol double dose group versus limicol simple dose group) | 4 weeks after baseline
Change from Baseline in blood total cholesterol, HDL-cholesterol and TAG levels after 4 weeks of supplementation (limicol double dose group versus limicol simple dose group versus placebo group) | 4 weeks after baseline
Change from Baseline in blood LDL-cholesterol, total cholesterol, HDL-cholesterol and TAG levels 4 weeks after end of supplementation (limicol double dose group versus limicol simple dose group versus placebo group) | 8 weeks after baseline
Change from Baseline in CK, LDH and other safety biomarkers levels after 4 weeks of supplementation (limicol double dose group versus placebo group versus placebo group) | 4 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Peltier, PhD, Study Director — Lescuyer Laboratory
Locations (1):
- Biofortis, Nantes, France

REFERENCES:
- [Derived] Barrat E, Zair Y, Sirvent P, Chauveau P, Maudet C, Housez B, Derbord E, Lescuyer JF, Bard JM, Cazaubiel M, Peltier SL. Effect on LDL-cholesterol of a large dose of a dietary supplement with plant extracts in subjects with untreated moderate hypercholesterolaemia: a randomised, double-blind, placebo-controlled study. Eur J Nutr. 2013 Dec;52(8):1843-52. doi: 10.1007/s00394-012-0486-2. Epub 2012 Dec 25. PMID 23266743